CLINICAL TRIAL: NCT06640257
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Trial Evaluating the Efficacy and Safety of SHR-1314 Injection in Adults With Active Psoriatic Arthritis
Brief Title: A Study of the Efficacy and Safety of SHR-1314 for Adult Active Psoriatic Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1314-308
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1314 injection (Experimental)
  Interventions: Drug: SHR-1314 injection
- placebo (Placebo Comparator)
  Interventions: Drug: SHR-1314 injection; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1314 injection — SHR-1314 injection
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This study is a randomized, double-blind, multicenter, placebo-controlled Phase III clinical study, consisting of a 4-week screening period, a 24-week core treatment period, a 24-week maintenance treatment period, and an 8-week safety follow-up period. It is planned to include 150 adult subjects with psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily signs an informed consent form before any procedures related to the research start;
2. At the time of screening, it met the 2006 psoriatic arthritis classification standard (CASPAR)；
3. There is active PsA before randomization;
4. Have active plaque psoriasis (at least one plaque skin lesion) at the time of screening, or have a history of plaque psoriasis;
5. Participants who have previously been treated with csDMARDs and/or NSAIDs still have active psoriatic arthritis disease.

Exclusion Criteria:

1. Existence of any of the following medical history or comorbid diseases: drug-induced psoriasis; other active inflammatory diseases or autoimmune diseases; history of organ transplantation; history of lymphocytic proliferation; severe infections, etc.
2. Have received psoriatic arthritis or psoriasis drugs, such as intra-articular injections, plant preparations, etc. within a certain period of time in the past.
3. Those who are allergic to the drug ingredients or excipients in this study, or are allergic to other biological agents.
4. A history of alcohol abuse or illegal drug abuse in pregnant or breastfeeding women, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving ACR 20 improvement at week 24 | Week 24

SECONDARY OUTCOMES:
The proportion of subjects who achieved ACR 50 improvement | Week 24
The proportion of subjects who achieved ACR 70 improvement | Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital of the Shanghai FuDan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided